CLINICAL TRIAL: NCT06837519
Title: A Randomized Double-Blind Trial Comparing Lidocaine and Dexmedetomidine Infusion and Their Combination on Perioperative Pain in Patients Undergoing Video-Assisted Thoracoscopic Surgery
Brief Title: Lidocaine and Dexmedetomidine Infusion and Their Combination on Perioperative Pain in Patients Undergoing Video-Assisted Thoracoscopic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sarah Ahmed, Lecturer of Anesthesia, Intensive care, and pain management, Faculty of Medicine, Ain Shams University, Cairo, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU R22/2025
Record Dates: First submitted 2025-02-15; First posted 2025-02-20 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Lidocaine; Dexmedetomidine; Infusion; Perioperative Pain; Video-Assisted Thoracoscopic Surgery
MeSH Terms: interventions — Lidocaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lidocaine group (Experimental): Patients will receive lidocaine 0.3 mg/kg over 10 min loading, 0.3 mg/kg/h infusion after induction of anesthesia as maintenance dose till 10 min before the end of the operation plus saline 0.9% with same rate of dexmedetomidine
  Interventions: Drug: Lidocaine
- Dexmedetomidine group (Experimental): Patients will receive dexmedetomidine 0.5 μg/kg infusion over 10 min as a loading dose then 0.5 μg/kg/h after induction of anesthesia as maintenance dose till 10 min before the end of the operation plus saline 0.9% with same rate of lidocaine.
  Interventions: Drug: Dexmedetomidine
- Lidocaine and Dexmedetomidine group (Experimental): Patients will receive lidocaine (0.3 mg/kg in 10 min loading, 0.3 mg/kg/h infusion) and dexmedetomidine infusions (0.5 μg/kg infusion over 10 min as a loading dose then 0.5 μg/kg/h) till 10 min before the end of the operation.
  Interventions: Drug: Lidocaine and Dexmedetomidine

INTERVENTIONS:
Drug: Lidocaine — Patients will receive lidocaine 0.3 mg/kg over 10 min loading, 0.3 mg/kg/h infusion after induction of anesthesia as maintenance dose till 10 min before the end of the operation plus saline 0.9% with same rate of dexmedetomidine.
  Arms: Lidocaine group
Drug: Dexmedetomidine — Patients will receive dexmedetomidine 0.5 μg/kg infusion over 10 min as a loading dose then 0.5 μg/kg/h after induction of anesthesia as maintenance dose till 10 min before the end of the operation plus saline 0.9% with same rate of lidocaine.
  Arms: Dexmedetomidine group
Drug: Lidocaine and Dexmedetomidine — Patients will receive lidocaine (0.3 mg/kg in 10 min loading, 0.3 mg/kg/h infusion) and dexmedetomidine infusions (0.5 μg/kg infusion over 10 min as a loading dose then 0.5 μg/kg/h) till 10 min before the end of the operation.
  Arms: Lidocaine and Dexmedetomidine group

SUMMARY:
This study aims to compare lidocaine and dexmedetomidine infusion and their combination on perioperative pain in patients undergoing video-assisted thoracoscopic surgery.

DETAILED DESCRIPTION:
Video-assisted thoracoscopic surgery (VATS) is a minimally invasive procedure allowing the reduction of surgical stress. However, postoperative pain management is crucial for patients undergoing VATS, as inadequate pain control can lead to complications (such as lung atelectasis), prolonged recovery, and decreased patient satisfaction.

Dexmedetomidine has shown positive effects on postoperative pain intensity, opioid consumption and other recovery parameters, such as postoperative nausea and vomiting (PONV), and speed of recovery.

Lidocaine has exhibited an excellent safety profile when administered as a low-dose infusion for cancer or non-cancer chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old.
* Both sexes.
* American Society of Anesthesiologists (ASA) physical status of I, II.
* Patients undergoing video-assisted thoracoscopic surgery (VATS) under general anesthesia.

Exclusion Criteria:

* Hypersensitivity to any of the used drugs.
* Coagulation disorder.
* Body mass index >35 kg/m2.
* History of chronic pain requiring daily opioids/steroids/clonidine/other α2 agonist/analgesics or any drugs acting on the central nervous system during the previous 2 weeks, and drug/alcohol abuse.
* Contraindication to the use of local anesthetics.
* Cardiovascular disease.
* Severe respiratory, renal or hepatic impairment.
* Insulin-dependent diabetes mellitus.
* Central nervous system or psychiatric disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Total morphine consumption | 24 hours postoperatively
  Rescue analgesia of morphine will be given as 3 mg bolus if the Visual Analogue Scale (VAS)> 3 to be repeated after 30 min if pain persists until the VAS < 4.

SECONDARY OUTCOMES:
Time of extubation | 24 hours postoperatively
  Time from the end of surgery till extubation
Time to the first request for the rescue analgesia | 24 hours postoperatively
  Time to the first request for the rescue analgesia (time from end of surgery to first dose of morphine administrated).
Degree of pain | 24 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the Visual Analogue Scale (VAS). VAS (0 represents "no pain" while 10 represents "the worst pain imaginable"). VAS will be assessed at 0, 4, 8, 12, 18 and 24h postoperatively.
Degree of patient satisfaction | 24 hours postoperatively
  The degree of patient satisfaction will be assessed on a 5-point Likert scale patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied).
Incidence of adverse events | 24 hours postoperatively
  Incidence of adverse events such as bradycardia, hypotension, nausea, vomiting, pruritis, respiratory depression, lidocaine toxicity (such as lightheadedness, somnolence, perioral numbness, dry mouth, metallic taste, dysarthria or fits) or any other complication will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.